CLINICAL TRIAL: NCT02899351
Title: The Evaluation of a Noninvasive Respiratory Monitor in Intubated Infants
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Viviane Nasr, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00023229
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Infants less than 12 months: intubated infants in ICU
  Interventions: Device: Respiratory Volume Monitor

INTERVENTIONS:
Device: Respiratory Volume Monitor
  Other Names: ExSpiron

SUMMARY:
In this research study, the investigators want to learn more about whether the Respiratory Volume Monitor (ExSpiron) can accurately measure breathing in infants less than 12 months of age. The Respiratory Volume Monitor uses up to 5 stickers that are placed on the chest to measure the amount of air going in and out of the lungs with each breath (Tidal Volume), the number of times per minute a breath is taken (Respiratory Rate), and the amount of air going in and out of the lungs per minute (Minute Ventilation).

It is important for medical staff to be able to collect information about breathing non-invasively because it may help determine if certain children are experiencing breathing problems sooner than the way it is currently detected.

The goal of this study is to determine if the Respiratory Volume Monitor works accurately in infants less than 12 months of age.

ELIGIBILITY:
Inclusion Criteria:

* less than 12 months of age
* currently intubated in the ICU

Exclusion Criteria:

* ExSpiron monitor will interfere with a healing surgical procedure site or standard of care

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Intubated infants less than 12 months of age who are admitted to an Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Respiratory rate accurately measured by the ExSpiron monitor during controlled ventilation | During 1 hour period in ICU
Tidal Volume accurately measured by the ExSpiron monitor during controlled ventilation | During 1 hour period in ICU
Minute ventilation accurately measured by the ExSpiron monitor during controlled ventilation | During 1 hour period in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Nasr, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Atkinson DB, Sens BA, Bernier RS, Gomez-Morad AD, Imsirovic J, Nasr VG. The Evaluation of a Noninvasive Respiratory Volume Monitor in Mechanically Ventilated Neonates and Infants. Anesth Analg. 2022 Jan 1;134(1):141-148. doi: 10.1213/ANE.0000000000005562. PMID 33929346